CLINICAL TRIAL: NCT03103737
Title: Evaluation of a Brief Psychological Intervention That Uses ICTs to Improve Well-being in Hospitalized Cancer Patients
Brief Title: Promotion of Emotional Well-being in Hospitalized Cancer Patients by Information and Communication Technologies (ICTs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rosa María Baños Rivera (Other)
Collaborators: Hospital Clínica Benidorm (Unknown); Universitat Jaume I (Other); Universitat Politècnica de València (Other)
Responsible Party: Sponsor-Investigator, Rosa María Baños Rivera, Full Professor, University of Valencia
Organization: University of Valencia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONCOTIC-II
Record Dates: First submitted 2017-03-22; First posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Cancer
Keywords: Well-being; Information and communication technologies; Hospital
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Psychological intervention composed by four sessions along 1 week. Participants can interact with virtual environments and a multimedia system for reminiscence purposes.
  Interventions: Behavioral: Virtual Reality (VR) and Reminiscence Intervention
- Control (No Intervention): Participants receive the medical treatment deliver by the hospital. After one week, they have the possibility to receive the psychological intervention.

INTERVENTIONS:
Behavioral: Virtual Reality (VR) and Reminiscence Intervention — First and third sessions are dedicated to remember positive and meaningful personal experiences. Second and fourth sessions are oriented to positive emotions by the use of VR. Participants can choose the virtual environment to work with.
  Arms: Intervention

SUMMARY:
The aim of this study is to test the efficacy of a brief psychological intervention composed by two therapeutic modules (virtual environments and reminiscence techniques) for the promotion of wellbeing of hospitalized adult cancer patients. Participants are randomly assigned to 2 conditions: intervention condition and control condition.

ELIGIBILITY:
Inclusion Criteria:

* adults with any cancer diagnosis
* hospitalized for at least 1 week
* Karnofsky functional state ≥50
* life expectancy ≥2 months

Exclusion Criteria:

* serious psychopathology
* cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-08-31 (Actual); Study Completion 2013-08-31 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983; adapted version of Tejero, Guimerá, Farré & Peri, 1986) | Change from baseline to 1 week
Fordyce Happiness Scale (Fordyce, 1988). | Change from baseline to 1 week

SECONDARY OUTCOMES:
Visual Analog Scale: Mood. | 4 days along 1 week
  Subjective mood change after each session.
Visual Analog Scale: Emotional State. Change pre-post sessions. | 4 days along 1 week
  positive affect, negative affect, well-being and calmness (5-point Likert scale)
Visual Analog Scale: Physical Discomfort. Change pre-post sessions. | 4 days along 1 week
  fatigue, pain and nausea-vomiting (5-point Likert scale)
Visual Analog Scale: Satisfaction with the Session | 4 days along 1 week
  pleasantness and perceived usefulness (5-point Likert scale)
Satisfaction with Intervention Scale (adapted version of Borkovec and Nau's, 1972). | 1 week
  satisfaction, recommendation, utility and discomfort (5-point Likert scale)
Distress Thermometer (Roth et al., 1998). | Change from baseline to 1 week
Time perception (based on Bayés et al., 1997). | 4 days along 1 week
  Participants has to indicate the session duration (in minutes). An objective measure of the time lapse is also registered by the researcher.